CLINICAL TRIAL: NCT07067671
Title: Evaluation of Regional Ventilation in Neuro-injured Patients Undergoing Weaning From Mechanical Ventilation
Brief Title: Regional Ventilation Evaluation During Neuro-injury Weaning Study
Acronym: ReVENtS
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250700; 2025-A01069-40 (Other: IDRCB)
Record Dates: First submitted 2025-06-13; First posted 2025-07-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acute Brain Injury; Mechanical Ventilation; Prolonged Weaning; Traumatic Brain Injury; Hypoxic-Ischemic Brain Injury; Intracerebral Hemorrhage
Keywords: Electrical Impedance Tomography; Ventilator Weaning; Neurocritical Care; ICU Monitoring; Spontaneous Breathing Trial; Extubation Failure; Respiratory Mechanics; PulmoVista; EIT; Brain-Injured Patients
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Hypoxia-Ischemia, Brain; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Internal Thoracic Impedance — Internal Thoracic Impedance is a non-invasive an imaging technique which use low alternative current through electrodes placed on a belt positioned at the level of the patient's rib cage. Images are constructed according to conductivity measured.

SUMMARY:
This study evaluates changes in regional lung ventilation using thoracic electrical impedance tomography (EIT) during the weaning process from mechanical ventilation in ICU patients with acute brain injury. It aims to identify predictive EIT patterns related to extubation outcomes.

DETAILED DESCRIPTION:
This is a prospective, single-center pilot study conducted in the intensive care unit. The study focuses on adult patients with acute brain injury requiring invasive mechanical ventilation for more than 48 hours. The aim is to assess regional alveolar ventilation using thoracic electrical impedance tomography (EIT) during different stages of ventilator weaning, including changes in ventilatory mode, spontaneous breathing trials, and, when feasible, around extubation or decannulation.

EIT provides dynamic, non-invasive real-time imaging of regional pulmonary ventilation. Data will be collected using a 16-electrode thoracic belt and analyzed retrospectively with dedicated software. The primary outcome measure is the Absolute Ventral-to-Dorsal Ventilation Difference, calculated from predefined regions of interest. Secondary outcomes include correlations with traditional ventilatory parameters (tidal volume, respiratory rate, oxygen saturation), end-expiratory impedance variation (ΔEELI), compliance changes, and extubation or decannulation failure defined by the need for reintubation within 7 days.

This study aims to improve understanding of regional ventilation patterns in brain-injured patients and assess the potential of EIT to predict weaning outcomes and guide personalized ventilatory strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Hospitalized in intensive care for an acute brain injury.
* Mechanical ventilation for more than 48 hours.
* Ventilator withdrawal planned in the next few days
* Social security coverage

Exclusion Criteria:

* Pregnancy
* Moribund patient / decision to stop treatment
* Patient under state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in intensive care for an acute brain injury under invasive mechanical ventilation for more than 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Absolute ventral-to-dorsal ventilation difference | From the start of the ventilator mode change or spontaneous breathing trial until 30 minutes after.
  The Absolute V-D Difference will be calculated as the average of the ventilation in the ventral regions (ROI1 and ROI2) minus the average of the ventilation in the dorsal regions (ROI3 and ROI4) during mechanical ventilation weaning. This outcome will provide insights into regional pulmonary ventilation distribution and its correlation with extubation outcomes.
  This difference is calculated as follows: (ROI_Value1 + ROI_Value2)/2 - (ROI_Value3 + ROI_Value4)/2 expressed as a percentage.

SECONDARY OUTCOMES:
Correlation between Absolute V-D Difference and Conventional Ventilatory Parameters | From the start of the ventilator mode change or spontaneous breathing trial until 30 minutes after
  This outcome will evaluate how the Absolute V-D Difference correlates with other monitoring parameters, such as tidal volume, respiratory rate, SpO₂, and end-tidal CO₂ (EtCO₂), throughout the weaning process.
End-Expiratory Lung Impedance (ΔEELI) | From 5 minutes before to 5 minutes after the 30-minute spontaneous breathing trial (i.e., total duration of 40 minutes)
  The monitoring of ΔEELI will be continuous throughout the spontaneous breathing trial, which lasts 30 minutes. Monitoring will begin at a stable baseline 5 minutes prior to the start of the trial and will continue until 5 minutes after its completion.
  Three specific time points will be collected and analyzed:
  1. EELI before the trial (baseline, 5 minutes prior),
  2. EELI at the end of the trial (30 minutes),
  3. EELI 5 minutes after resumption of mechanical ventilation
Correlation between ΔEELI and Extubation/Decannulation Failure | 7 days post-extubation or post-deventilation.
  This secondary outcome assesses the relationship between changes in end-expiratory impedance (ΔEELI) and extubation or decannulation failure, defined as reintubation or need for reventilation within 7 days.
Pulmonary Compliance Variation during Ventilator Changes and Spontaneous Breathing Trials | From the start of ventilator mode change or spontaneous breathing trial until 30 minutes after.
  This measure will track the changes in regional pulmonary compliance in response to adjustments in ventilator parameters (e.g., PEEP, tidal volume) and spontaneous breathing trials.
Absolute V-D Difference and Extubation Failure | 7 days post-extubation or post-deventilation.
  This outcome will examine the correlation between the Absolute V-D Difference and extubation failure, defined as reintubation or the need for reventilation within 7 days post-extubation or post-deventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Gaugain, MD, Principal Investigator — APHP
Locations (1):
- Hôpital Lariboisière - APHP, Paris, France, France

IPD SHARING:
Plan to Share IPD: No